CLINICAL TRIAL: NCT03040752
Title: Comparative Study Between Nifedipine and Ritodrine as Maintenance Tocolytic Therapy in Preterm Labor: A Randomized Controlled Trial
Brief Title: Comparative Study Between Nifedipine and Ritodrine as Maintenance Tocolytic Therapy in Preterm Labor
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed M Maged, MD, Assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 157
Record Dates: First submitted 2017-01-31; First posted 2017-02-02 (Estimated); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth | interventions — Nifedipine; Ritodrine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nifedipine (Active Comparator): nifedipine 20 mg tablets (Epilat Retard®, EIPICO, Egypt) twice daily, starting 12 hours after arrest of threatened preterm labor
  Interventions: Drug: Nifedipine 20 Mg
- Ritodrine (Active Comparator): Ritodrine 5 mg tablets (Yutopar®, PHARCO, Alexandria) every 6 hours, starting 12 hours after arrest of threatened preterm labor.
  Interventions: Drug: Ritodrine Oral Tablet

INTERVENTIONS:
Drug: Nifedipine 20 Mg — nifedipine 20 mg tablets (Epilat Retard®, EIPICO, Egypt) twice daily, starting 12 hours after arrest of threatened preterm labor
  Other Names: Epilate retard
  Arms: Nifedipine
Drug: Ritodrine Oral Tablet — Ritodrine 5 mg tablets (Yutopar®, PHARCO, Alexandria) every 6 hours, starting 12 hours after arrest of threatened preterm labor
  Other Names: Yutopar
  Arms: Ritodrine

SUMMARY:
A randomized controlled double blinded study included 200 women with preterm contractions. After successful arrest of contractions women were randomized into 2 equal groups: GI women received nifedipine 20 mg tablets twice daily and GII women received Ritodrine 5 mg tablets every 6 hours. The primary outcome was gestational age at delivery and the secondary outcomes include episodes of recurrent preterm labor, mode of delivery, maternal side effects and neonatal outcome

DETAILED DESCRIPTION:
Women included in the study were diagnosed as preterm labor defined according to American Academy of Pediatrics and the American College of Obstetricians and Gynecologists (2012) with regular contractions before 37 weeks that are associated with cervical change [12].

Regular uterine contractions means at least 4 in 20 minutes or 8 in 60 minutes) and cervical changes are either cervical dilation more than 1 cm, and/or cervical effacement ≥ 80%. Threatened preterm labour was defined as contractions without any appreciable cervical changes. Women included were between 18 and 40 years old at gestational age between 28 and 34 weeks. Women with failed tocolytic treatment to stop uterine contractions, those with established preterm labor (cervical dilatation ≥ 4 cm), with multifetal pregnancy, fetal anomalies or those with contraindication of continuation of pregnancy (antepartum hemorrhage, premature rupture of membranes, evidence of intrauterine infections or non reassuring fetal heart rate tracing) were excluded from the study.

During the pre-selection visit, exclusion and inclusion criteria were applied; with recording of full medical history, findings on abdominal ,local and ultrasound examination.

When the patient's consent was obtained, digital vaginal examination was done prior to start of medication Treatment of TPL was achieved through Indomethacin administered rectally. A dose of 50 to 100 mg is followed at 8-hour intervals not to exceed a total 24-hour dose of 200 mg for a maximum of 48 hours [4].

After successful arrest of contractions women were randomized using automated web based randomization system ensuring allocation concealment into 2 equal groups: GI women received nifedipine 20 mg tablets (Epilat Retard®, EIPICO, Egypt) twice daily, starting 12 hours after arrest of threatened preterm labor(The cost is 20 tab=5.20 LE) and GII women received Ritodrine 5 mg tablets (Yutopar®, PHARCO, Alexandria) every 6 hours, starting 12 hours after arrest of threatened preterm labor.(The cost is 20 tab=20LE Treatment was maintained till 37 weeks of gestation unless established preterm delivery commence

ELIGIBILITY:
Inclusion Criteria:

* Women included in the study were diagnosed as preterm labor defined according to American Academy of Pediatrics and the American College of Obstetricians and Gynecologists (2012) with regular contractions before 37 weeks that are associated with cervical change .

Regular uterine contractions means at least 4 in 20 minutes or 8 in 60 minutes) and cervical changes are either cervical dilation more than 1 cm, and/or cervical effacement ≥ 80%. Threatened preterm labour was defined as contractions without any appreciable cervical changes. Women included were between 18 and 40 years old at gestational age between 28 and 34 weeks

Exclusion Criteria:

* Women with failed tocolytic treatment to stop uterine contractions,
* those with established preterm labor (cervical dilatation ≥ 4 cm),
* multifetal pregnancy
* fetal anomalies
* those with contraindication of continuation of pregnancy (antepartum hemorrhage, premature rupture of membranes, evidence of intrauterine infections or non reassuring fetal heart rate tracing)

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 200 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
gestational age at delivery | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, Principal Investigator — Kasr Alainy medical school
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wilson A, Hodgetts-Morton VA, Marson EJ, Markland AD, Larkai E, Papadopoulou A, Coomarasamy A, Tobias A, Chou D, Oladapo OT, Price MJ, Morris K, Gallos ID. Tocolytics for delaying preterm birth: a network meta-analysis (0924). Cochrane Database Syst Rev. 2022 Aug 10;8(8):CD014978. doi: 10.1002/14651858.CD014978.pub2. PMID 35947046